CLINICAL TRIAL: NCT01643629
Title: A Prospective Multicentric Open Label Randomized Bio-Interventional Phase I/II Pilot Study To Evaluate The Safety And Efficacy Of Autologous Human Platelet Lysate (HPL) For Treatment Of Androgenetic Alopecia (AGA)
Brief Title: A Study to Determine the Safety and Efficacy of Autologous Human Platelet Lysate for Treatment of Androgenetic Alopecia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/HPL-AGA/11-12/001A
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study arm A (Other): Study arm A will include subjects receiving three doses of Autologous Human Platelet Lysate at an interval of one month each.
  Interventions: Biological: Autologous Human Platelet Lysate (HPL)
- Control Arm B (Other): Control arm B will include subjects receiving Standard therapy
  Interventions: Other: 2 % Minoxidil and /or Finasteride

INTERVENTIONS:
Biological: Autologous Human Platelet Lysate (HPL) — Study arm A will include subjects receiving three doses of Autologous Human Platelet Lysate at an interval of one month each.
  Arms: Study arm A
Other: 2 % Minoxidil and /or Finasteride — Control arm B subjects will receive Standard therapy (2% Minoxidil and/or Finasteride)
  Arms: Control Arm B

SUMMARY:
This is a multicentre, open label, randomized, pilot study to evaluate safety and efficacy of Human Platelet Lysate (HPL) in subjects with Androgenetic Alopecia. The study is being conducted at 2 centers in India. The primary endpoints are Improvement in Caliber & Density of hair and Improvement in Photographic assessment from randomization to end of study. The secondary endpoints are Physicians and Patients self assessment score.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged between 18 to 50 years (both inclusive) and in general good health
* Subjects willing to refrain from other AGA treatments during the entire study duration
* Subjects who are willing to give informed consent and adhere to the study protocol.

Exclusion Criteria:

* Subjects aged <18 or > 50 years
* Subjects with dermatological disorder of scalp that might interfere with study evaluation
* Subjects on Anti-coagulant therapy
* Subjects with clinically significant medical or psychiatric disease as determined by the investigator.
* Subjects with dermatological disorder of scalp that might interfere with study evaluation
* Subjects unwilling to or unable to comply with the study protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Change in Calibre & Density of Hair as assessed by Folliscope | Day 0, Month 4, End of study - Month 6

SECONDARY OUTCOMES:
Photographic Assessment | Day 0, Month1, Month 2, Month 3, Month 4, Month 5, Month 6

OTHER OUTCOMES:
Physician's Assessment Score | End of study - Month 6
Patient's Assessment Score | End of study - Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Rajendarsingh Rajput, Dr., Principal Investigator — Dr. Rajesh Rajput Hair Restore; Sandeep Sattur, Dr., Principal Investigator — Hairrevive
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India